CLINICAL TRIAL: NCT01407237
Title: Physiologic Investigation of the Renin Angiotensin Aldosterone Axis in HIV
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2011P000250
Record Dates: First submitted 2011-07-27; First posted 2011-08-02 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: HIV-infection
Keywords: HIV-infection; renin; aldosterone; visceral fat
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- HIV-infected Individuals
  Interventions: Drug: Angiotensin II Infusion
- non-HIV-infected Individuals
  Interventions: Drug: Angiotensin II Infusion

INTERVENTIONS:
Drug: Angiotensin II Infusion — Angiotensin II (Bachem) will be infused at 0.3 ng/kg/min for 30 minutes, then 1.0 ng/kg/min for 30 minutes, then 3.0 ng/kg/min for 30 minutes; at baseline and at each infusion concentration, serum aldosterone will be measured. BP and heart rate will be monitored at baseline and every 2 minutes during the infusion.

SUMMARY:
The purpose of this study is to see if individuals with HIV-infection, particularly those with increased belly fat, have abnormalities in the renin angiotensin aldosterone axis. Renin, angiotensin, and aldosterone are hormones that regulate salt and water balance in the body, and they may also have effects on sugar metabolism and cardiovascular health. There is some evidence that individuals with HIV-associated abdominal fat accumulation may have increased aldosterone, which may contribute to abnormalities in sugar metabolism and increased cardiovascular disease seen in HIV. The purpose of this study is the measure renin, angiotensin, and aldosterone activity, as well as other hormonal axes, in people with and without HIV infection, and with and without increased belly fat. The investigators hypothesize that aldosterone will be increased in HIV-infected individuals compared to those without HIV-infection, and that aldosterone will be further increased in HIV-infected individuals with increased abdominal fat compared to those without abdominal fat accumulation.

ELIGIBILITY:
Inclusion Criteria:

1. Stable use of antiretroviral therapy for at least 3 months (HIV group)
2. Age ≥ 18 and ≤ 65 years of age

Exclusion Criteria:

1. Antihypertensive use, including angiotensin converting enzyme inhibitors or angiotensin II receptor blocker use, diuretics, beta-blockers, calcium-channel blockers, potassium supplements, and spironolactone; and/or blood pressure (BP) >140/90 at screen
2. Current or recent steroid use within last 2 months.
3. Known diabetes and/or use of antidiabetic medications
4. Creatinine > 1.5 mg/dL
5. Potassium (K) > 5.5 mEq/L
6. Hemoglobin (Hgb) < 11.0 mg/dL
7. Alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN)
8. Thyroid disease/abnormal thyroid stimulating hormone (TSH)
9. Significant electrocardiographic abnormalities at screen such as heart block or ischemia
10. History of congestive heart failure, stroke, myocardial infarction, or known coronary artery disease (CAD)
11. For women: Pregnant or actively seeking pregnancy, or breastfeeding
12. Estrogen, progestational derivative, growth hormone (GH), growth hormone releasing hormone (GHRH) or ketoconazole use within 3 months.
13. Current viral, bacterial or other infections (excluding HIV)
14. Current cigarette smoker/use of nicotine (patch/gum) or current active substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 HIV-infected and 50 non-HIV-infected male and female volunteers, ages 18-65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
24-hour urine aldosterone to creatinine ratio | baseline

SECONDARY OUTCOMES:
Plasma Renin Activity | baseline
Aldosterone response to Angiotensin II Infusion | baseline
Flow mediated dilation | baseline
Intramyocellular Lipid | baseline
Hepatic fat | baseline
Insulin stimulated glucose uptake | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bogorodskaya M, Fitch KV, Burdo TH, Maehler P, Easly RM, Murray GR, Feldpausch M, Adler GK, Grinspoon SK, Srinivasa S. Serum Lipocalin 2 (Neutrophil Gelatinase-Associated Lipocalin) in Relation to Biomarkers of Inflammation and Cardiac Stretch During Activation of the Renin-Angiotensin-Aldosterone System in Human Immunodeficiency Virus. J Infect Dis. 2019 Sep 26;220(9):1420-1424. doi: 10.1093/infdis/jiz346. PMID 31298286
- [Derived] Murphy CA, Fitch KV, Feldpausch M, Maehler P, Wong K, Torriani M, Adler GK, Grinspoon SK, Srinivasa S. Excessive Adiposity and Metabolic Dysfunction Relate to Reduced Natriuretic Peptide During RAAS Activation in HIV. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1558-1565. doi: 10.1210/jc.2017-02198. PMID 29408981
- [Derived] O'Malley TK, Burdo TH, Robinson JA, Fitch KV, Grinspoon SK, Srinivasa S. Acute hyperinsulinemia effects on systemic markers of immune activation in HIV. AIDS. 2017 Jul 31;31(12):1771-1773. doi: 10.1097/QAD.0000000000001545. PMID 28514281
- [Derived] Srinivasa S, Burdo TH, Williams KC, Mitten EK, Wong K, Fitch KV, Stanley T, Adler GK, Grinspoon SK. Effects of Sodium Restriction on Activation of the Renin-Angiotensin-Aldosterone System and Immune Indices During HIV Infection. J Infect Dis. 2016 Nov 1;214(9):1336-1340. doi: 10.1093/infdis/jiw392. Epub 2016 Aug 22. PMID 27549584
- [Derived] Srinivasa S, Fitch KV, Wong K, Torriani M, Mayhew C, Stanley T, Lo J, Adler GK, Grinspoon SK. RAAS Activation Is Associated With Visceral Adiposity and Insulin Resistance Among HIV-infected Patients. J Clin Endocrinol Metab. 2015 Aug;100(8):2873-82. doi: 10.1210/jc.2015-1461. Epub 2015 Jun 18. PMID 26086328